CLINICAL TRIAL: NCT01846026
Title: Immunomodulating and Clinical Effects of Vitamin D on Remission Induction in Patients With Moderate and Severe Ulcerative Colitis, Undergoing Treatment With Infliximab.
Brief Title: Ulcerative Colitis and Vitamin D Supplementation
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: At the planned study start new treatment guidelines for this disease with new drugs were implemented in clinical practice.
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009/1392-13 (REK); 2009-015649-21 (EudraCT Number)
Record Dates: First submitted 2013-04-30; First posted 2013-05-03 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-06

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D (Experimental): Decristol (cholecalciferol) 20000 IU per capsule
  1 capsule per week
  Interventions: Drug: Vitamin D
- Placebo (Placebo Comparator): capsule with peanut oil
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Vitamin D — compare how vitamin D influences the course of ulcerative colitis versus placebo
  Other Names: Cholecalciferol
  Arms: Vitamin D
Drug: placebo
  Arms: Placebo

SUMMARY:
Ulcerative colitis (UC) is an inflammatory disease involving the colonic mucosa, with bleedings and ulcerations. Consequences are destroyed mucosal barrier and increased permeability. Several cytokines are described to mediate the progressive course of ulcerative colitis and it is considered nowadays an immunologic disease. Patients with UC have often low levels of vitamin D and elevated prevalence of osteoporosis.

In vitro studies demonstrate that vitamin D has an immunomodulating effect, and may have a direct healing action on colonic mucosa has been described in animal studies. One can therefore rise a hypothesis that vitamin D supplementation could be crucial in patients with UC. To our knowledge, it has not been performed randomized clinical trials to study these possible effects of vitamin D and it has not been studied the effects of vitamin D on the relapse frequency and immunological composition of colic mucosa in patient with moderate to severe ulcerative colitis.

Objectives for our study are as follows: To examine if high-dose vitamin D supplementation in patients with moderate to severe ulcerative colitis:

* reduces relapse frequency and increase the duration of the Infliximab induced remission
* mediates and changes the cytokines composition in the colic mucosa
* decreases the excretion of calprotectin in feces and reduces the concentration of inflammation markers
* augments bone mass

ELIGIBILITY:
Inclusion Criteria:

* Men and women older than18 years old, diagnosed with UC (either debut or relapsed chronic UC), moderate or severe, where it is an indication to treat with infliximab.

Exclusion Criteria:

* Primary hyperparathyroidism (PHPT)
* Sarcoidosis
* Renal failure (serum creatinine > 125 mumol/L in men or > 105 mumol/L in women)
* Those, who use solarium routinely are not included
* Pregnant or breastfeeding women, otherwise women of fertile age must be on approved birth control methods during the study
* Renal stones last 15 years
* Cancer of any origin, diagnosed during last 5 years
* Unstable angina pectoris

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2014-04 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
number of patients with remission | 12 months after start of intervention
  Mandatory criterion of remission: clinical remission (defined as Mayo score <= 1, including endoscopic findings) and non-mandatory: laboratory (calprotectin < 100, WBC and SR within reference range). These criteria will be assessed at 12 month after the start of intervention

SECONDARY OUTCOMES:
change in fecal calprotectin | 12 months after start of intervention
  change in fecal calprotectin compared to baseline value
change in bone mineral density (whole body) | 12 months after the start of intervention
  change in bone mineral density in whole body, measured with DEXA (t-score and z-score)
change in fecal calprotectin | 3 months
  change in fecal calprotectin
change in tnf-alpha levels in colonic mucosa | 3 months
  change in mucosal tnf-alpha levels. Biopsies will be taken with the forceps from the colonic mucosa (colon sigmoid) and stored in RNA later media for the further analysis for TNF alpha concentration with PCR method.
change in tnf-alpha (in colonic mucosa) | 12 months after baseline
  Biopsies and analysis will be carried out as described ata 3 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Elena Kamycheva, MD, PhD, Principal Investigator — Medical Clinic, University Hospital of North Norway
Locations (1):
- University Hospital of North Norway, Tromsø, Norway